CLINICAL TRIAL: NCT05561478
Title: Comparison of Visual Outcomes After Implantation of the Synthesis Plus and Synthesis Plus Toric
Acronym: DETPLUST
Status: Recruiting | Type: Observational
Sponsor: Cutting Edge SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02415-36
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-09

CONDITIONS: Cataract; Surgery; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Test device (Synthesis Plus Toric): Requiring bilateral cataract surgery with pre-existing astigmatism
  Interventions: Device: Implantation of Synthesis Plus Toric IOL (investigational device)
- Control device (Synthesis Plus): Requiring bilateral cataract surgery
  Interventions: Device: Implantation of Synthesis Plus IOL (control device)

INTERVENTIONS:
Device: Implantation of Synthesis Plus IOL (control device) — Synthesis Plus IOLs are indicated for primary implantation for the visual correction of aphakia in adult patients.
  Groups: Control device (Synthesis Plus)
Device: Implantation of Synthesis Plus Toric IOL (investigational device) — Synthesis Plus Toric IOLs are indicated for primary implantation for the visual correction of aphakia in adult patients with pre-existing astigmatism.
  Groups: Test device (Synthesis Plus Toric)

SUMMARY:
Prospective controlled monocentric study to determine the non-inferiority of the distance-corrected intermediate visual acuity at 66 cm of the SYNTHESIS PLUS TORIC with respect to the SYNTHESIS PLUS IOL.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 50 years old
* Patient requiring bilateral cataract surgery
* Regular corneal astigmatism >0.5D measured by MS-39 (SimK keratometry and regularity determined by the topography) for patients implanted with SYNTHESIS PLUS TORIC or Regular corneal astigmatism lower or equal to 0.5 D dioptres by MS-39 (SimK keratometry and regularity determined by the topography) for patients implanted with SYNTHESIS PLUS.
* Expected postoperative astigmatism ≤ 0.75D diopter
* Corneal astigmatism ≤4D
* IOL spherical equivalent power requested between 15D and 25D
* Signed informed consent
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures

Non inclusion Criteria:

* Patients with a potential postoperative visual acuity of less than 5/10, in particular due to degenerative visual disorders, poor retinal function or a damaged cornea.
* Amblyopia with a visual acuity potential of less than 5/10
* IOL power needed outside the spherical equivalent diopter range: 15 to 25D
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Irregular astigmatism
* Subject with postoperative astigmatism, expected > 0.75 D.
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Patients with chronic uveitis
* Pupil abnormalitis (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions, diameter (pupil>4mm or <2.5 mm in photopic conditions))
* Narrow anterior chambers (ACD ≤ 2.5 mm)
* Any corneal pathology potentially affecting the topography (eg. Keratoconus),
* Monophthalma patients
* Phacodonesis

Exclusion criteria:

* Complicated surgery
* Inability to place the intraocular lens safely at the location planned
* Subjects with zonular laxity
* Postoperative endophthalmitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring bilateral cataract surgery
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
DCIVA at 66 cm | 1 month
  The primary objective of this study is to determine the non-inferiority of the distance-corrected intermediate visual acuity at 66 cm of the SYNTHESIS PLUS TORIC with respect to the SYNTHESIS PLUS

SECONDARY OUTCOMES:
Monocular UDVA | 1 month
  distance
Monocular BCDVA | 1 month
  distance
Monocular UIVA | 1 month
  66 cm
Monocular DCIVA | 1 month
  66 cm
Refraction | 1 month
  subjective
Potential complications | 1 month
  postoperative
Rotational stability | Peroperatively, day 0, Month 1
  in degrees
Subjective quality of vision | 1 month
  PROM

CONTACTS AND LOCATIONS:
Overall Officials: Boris Dethinne, MD, Principal Investigator — Visis
Locations (1):
- VISIS, Perpignan, France